CLINICAL TRIAL: NCT01150175
Title: Double-blind Placebo Controlled Trial on Direct Endomyocardial Injection of Autologous Bone Marrow Cells for Enhancement of Neovascularization in Patients With Ischaemic Heart Failure (END-HF)
Brief Title: Direct Endomyocardial Injection of Autologous Bone Marrow Cells to Treat Ischaemic Heart Failure
Acronym: END-HF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Prof. HF TSE, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HKCTR-763; END-HF Version 1:17-5-08
Record Dates: First submitted 2010-05-24; First posted 2010-06-24 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2010-06

CONDITIONS: Coronary Artery Disease
Keywords: END-HF
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous bone marrow cells (Experimental)
  Interventions: Procedure: Endomyocardial Injection of Autologous Bone Marrow Cells
- Plasma (Placebo Comparator)
  Interventions: Procedure: Endomyocardial Injection of Plasma

INTERVENTIONS:
Procedure: Endomyocardial Injection of Autologous Bone Marrow Cells — Endomyocardial Injection of Autologous Bone Marrow Cells
  Other Names: END-HF
  Arms: Autologous bone marrow cells
Procedure: Endomyocardial Injection of Plasma — Endomyocardial Injection of Plasma
  Other Names: END-HF
  Arms: Plasma

SUMMARY:
The purpose of this study is to determine whether direct endomyocardial injection of autologous bone marrow cells is effective for enhancement of neovascularisation in patients with ischaemic heart failure.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) remains to be one of the leading causes of mortality and morbidity worldwide. Despite the optimal use of anti-anginal medications and coronary revascularization, a large number of patients with CAD suffer from severe symptoms with disabling angina and heart failure (HF). Experimental and pilot clinical studies provided evidence of the safety and potential efficacy of a strategy of intramyocardial transplantation of autologous bone marrow (BM) cells for neovascularisation of chronically ischemic myocardium. Nevertheless, the possible potent placebo effect on symptoms observed in these pilot studies highlights the need for a randomized, placebo-controlled group to prove the clinical efficacy of cell based angiogenic therapy for treatment of severe CAD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old
* Canadian cardiovascular (CV) Class II-IV angina and/or NYHA class II-III HF symptoms
* Received stable and "best" cardiac medical therapy including long-acting nitrates, beta-blocker, and angiotensin-converting enzyme inhibitors without control of symptoms.
* Not suitable for conventional revascularization by their referring cardiologist.
* LVEF <40% by echocardiography.
* Recent coronary angiogram (within the last 6 months) to document the coronary anatomy and insure the presence of CAD that is not amenable to standard revascularization procedures.
* creatinine less than 250mmol/L, normal liver function, and normal blood count: WBC, granulocytes; platelet count, Hb.
* Reversible perfusion defect on single photon emission computed tomography (SPECT)
* Able to walk on treadmill
* Hemodynamically stable
* Subject is willing to comply with specified follow-up evaluations.
* All patients give written informed consent.

Exclusion Criteria:

* Atrial fibrillation
* History of syncope or major ventricular arrhythmias such as sustained ventricular tachycardia or ventricular fibrillation
* Severe valve disease
* Aortic or mitral valve prosthesis
* History of cancer in last 5 years
* Acute or chronic active sepsis, including HIV positive; hepatitis B or C positive
* Left ventricular wall thickness less than 8 mm in the target territory
* Left ventricular thrombus and/or spontaneous echo-contrast in the LV detected by echocardiography or LV aneurysm
* Severe aorto-femoral-iliac disease
* Recent heart attack within the last 30 days
* Hypertrophic or restrictive cardiomyopathy
* Severe co-morbidity associated with a reduction in life expectancy of less than 1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-07; Primary Completion 2011-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
MRI ejection fraction | MRI ejection fraction changed from baseline to 6 months

SECONDARY OUTCOMES:
Changes in exercise duration and MVO2 using standardized treadmill testing(modified Bruce protocol) from baseline to 6 months | Baseline to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. HF Tse, Hong Kong, China